CLINICAL TRIAL: NCT02493712
Title: A Phase 2a, Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Trial of IBD98-M Delayed-release Capsules to Induce Remission in Patients With Active, Mild to Moderate Ulcerative Colitis
Brief Title: A Phase 2a, Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Trial of IBD98-M
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Holy Stone Healthcare Co., Ltd (Industry)
Collaborators: inVentiv Health Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBD98-M-2002
Record Dates: First submitted 2015-07-07; First posted 2015-07-09 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- High dose (Experimental): High dose, twice a day for 6 weeks.
  Interventions: Drug: High dose
- Placebo: C (Placebo Comparator): Placebo, twice a day
  Interventions: Drug: Placebo
- Low dose (Experimental): Low dose, twice a day for 6 weeks
  Interventions: Drug: Low dose

INTERVENTIONS:
Drug: High dose — 6 capsules of IBD98-M, twice a day
  Other Names: Mesalamine-Sodium Hyaluronic 200 mg-23 mg
  Arms: High dose
Drug: Low dose — 4 capsules of IBD98-M
  Other Names: Mesalamine-Sodium Hyaluronic 200 mg-23 mg
  Arms: Low dose
Drug: Placebo — Placebo
  Arms: Placebo: C

SUMMARY:
IBD98-M-2002 is a phase 2a , Randomized, Double blind, Placebo-controlled of IBD98-M Delayed Release capsules in subjects with Mild to Moderately Ulcerative Colitis to investigate the clinical efficacy of IBD98-M delayed release capsules (in a fixed combination) over a 6-week treatment period and 2 weeks follow up.

DETAILED DESCRIPTION:
Study IBD98-M-2002 is a Phase 2a, multicenter, randomized, double-blind, parallel-group, placebo-controlled study in patients with active, mild to moderate UC. It is being conducted as an exploratory proof of concept study to investigate the clinical efficacy of IBD98-M delayed-release capsules (in a fixed combination) over a 6-week treatment period and a 2-week follow-up period.

Patients will be screened for study enrollment up to 4 weeks prior to randomization (Visit 3). During the screening period, patients will be evaluated by conducting laboratory tests, physical examination, and sigmoidoscopy. To be eligible, patients are to have a score of ≥4 and ≤10 on the UCDAI, and a score of ≥1 on the UCDAI endoscopy subscore. In addition, the diagnosis of UC must be confirmed by endoscopic and histologic evidence in the past; if prior confirmation is not available, this must be done at the time of screening endoscopy. After the screening visits, eligible patients will be randomized to 1 of 3 study groups: (1) IBD98 M 0.8 g/day (mesalamine 0.8 g with sodium hyaluronate 92 mg), (2) IBD98 M 1.2 g/day (mesalamine 1.2 g with sodium hyaluronate 138 mg), or (3) placebo. Up to 51 patients will be enrolled in this study (including drop-out patients), with 17 patients randomized to each treatment group. Patients will be encouraged to take their medication at the same time every day.

During the study, patients will visit the clinic on 7 occasions: 2 visits during the screening period (the second screening visit is the baseline visit); 4 visits during the treatment period, Visits 3, 4, 5, and 6/early termination at Weeks 0, 2, 4, and 6; and 1 visit at the end of the follow-up period, Visit 7 at Week 8. Patients will record the dates/times of dosing (after randomization), concomitant medication, and symptoms and adverse events (AEs) in a daily diary starting at Visit 1 and continuing until the end of treatment (Visit 6/early termination). Rescue medication will not be permitted during the 6 weeks of the treatment period, and patients who are considered to not be benefiting from the therapy can be withdrawn and assigned an appropriate alternative UC treatment by the Investigator. Compliance will be assessed throughout the study by determining the amount of unused medication. Records will be kept of all medication dispensed, used, and returned by each patient. At the end of the study, all unused trial medication and used packaging will be returned to the Sponsor. All study medication will be accounted for and any discrepancies documented.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 and <75 years, suffering from UC for at least 6 months prior to screening
2. Female patients must be postmenopausal, sterile, or have a negative urine pregnancy test prior to entering the study and use adequate contraception during the study if of childbearing potential.
3. Diagnosis of active UC with UCDAI ≥4 and ≤10, with endoscopy score of ≥1 in the UCDAI mucosal appearance subscore

Exclusion Criteria:

1. Patients diagnosed with Crohn's disease, indeterminate colitis, or ischemic colitis
2. Female patients who are pregnant or breastfeeding
3. Ulcerative proctitis with ≤15 cm of disease
4. Patients with infectious colitis as determined by assessment for Clostridium difficile (C. difficile) and fecal pathogens at screening or treatment for C. difficile within 30 days prior to screening
5. History of or current evidence of toxic megacolon, fulminant colitis (e.g., Lichtiger score of ≥10), colonic perforation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-01; Primary Completion 2018-07 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Danese, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Milan, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Started recruitment on 2016/01/01 Completed recruitment on 2018/07/01
Pre-assignment Details: No patient was excluded before assignment to groups.
Period: Overall Study
Arm/Group | High Dose | Placebo: C | Low Dose
Started | 16 | 18 | 17
Completed | 14 | 12 | 11
Not Completed | 2 | 6 | 6
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 5 | 3

BASELINE CHARACTERISTICS:
Population: All enrolled patients were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose | Placebo: C | Low Dose | Total
Number analyzed (Participants) | 16 | 18 | 17 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 17 | 49
  >=65 years | 1 | 1 | 0 | 2
Age, Continuous [Median (Full Range); unit: years] | 43.5 [22 to 69] | 47.5 [21 to 69] | 35 [20 to 54] | 45 [20 to 69]
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (12.23) | 45.8 (12.21) | 36.6 (10.68) | 41.9 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 5 | 23
  Male | 7 | 9 | 12 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 16 | 17 | 15 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 16 | 17 | 15 | 48
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] | 16 | 18 | 17 | 51
Region of Enrollment [Number; unit: participants]
  Italy | 16 | 18 | 17 | 51
UC remission [Count of Participants; unit: Participants] — remission was defined as having a modified Ulcerative Colitis Disease Activity Index [UCDAI] score of ≤1, with a score of 0 for rectal bleeding and stool frequency, no mucosal friability, and a sigmoidoscopy score not exceeding 1
  Participants | 16 | 18 | 17 | 51

OUTCOME MEASURES:

1. Primary Outcome: Remission Rate
Description: Percentage of patients in remission over a 6-week treatment period. Remission is defined as a modified UCDAI (Ulcerative Colitis Disease Activity Index) score of ≤1, with a score of 0 for rectal bleeding and stool frequency, no mucosal friability, and sigmoidoscopy score not exceeding 1).
  Modified UCDAI scoring system is sum of following 4 subscores (parameters). Higher score means worst disease condition.
  Rectal bleeding: score 1 (Streaks of blood), score 2 (obvious blood), score 3 (Mostly Blood) Stool frequency: score 1 (1-2/day> normal), score 2 (3-4/day >normal), score 3 (>4/day> normal) Mucosal appearance: score 1 (Erythema, decreased vascular pattern, Minimal granularity), score 2 (Marked erythema, Friability, Granularity, Absent vascular pattern, Bleeding minimal trauma, No ulcerations), score 3 (Ulceration Spontaneous bleeding) Physician's Global Assessment: score 1 (mild), score 2 (Moderate), score 3 (Severe)
Time Frame: 6 weeks
Population: The percentage of patients in remission at Week 6 is summarized for the ITT population.
Measure: Count of Participants; unit: Participants
Groups:
- High Dose Group: IBD98-M 1.2 g/day group
- Low Dose Group: IBD98-M 0.8 g/day group
- Placebo: Placebo capsule, 6 capsules/day
Arm/Group | High Dose Group | Low Dose Group | Placebo
Number analyzed (Participants) | 16 | 17 | 18
Participants | 2 | 1 | 2

2. Secondary Outcome: Improvement Rate
Description: Clinical improvement over a 6-weeks treatment period was defined as a ≥ 3 point reduction from Baseline in the modified UCDAI (Ulcerative Colitis Disease Activity Index ) score.
  Modified UCDAI scoring system is sum of following 4 subscores (parameters). Higher score means worst disease condition.
  Rectal bleeding: score 1 (Streaks of blood), score 2 (obvious blood), score 3 (Mostly Blood) Stool frequency: score 1 (1-2/day> normal), score 2 (3-4/day >normal), score 3 (>4/day> normal) Mucosal appearance: score 1 (Erythema, decrased vascular pattern, Minimal granularity), score 2 (Marked erythema, Friability, Granularity, Absent vascular pattern, Bleeding minimal trauma, No ulcerations), score 3 (Ulceration Spontaneous bleeding) Physician's Global Assessment: score 1 (mild), score 2 (Moderate), score 3 (Severe)
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Group | Low Dose Group | Placebo
Number analyzed (Participants) | 16 | 17 | 18
Participants | 5 | 3 | 3

ADVERSE EVENTS:
Time Frame: up to 8 weeks - 6 weeks treatment and 2 weeks follow-up
Description: The gastro disorder is not the high risk for mortality
Arm/Group | High Dose Group | Low Dose Group | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 1/18
Other Adverse Events (participants affected / at risk) | 6/16 | 8/17 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Group (N=16) | Low Dose Group (N=17) | Placebo (N=18)
WORSENING OF ULCERATIVE COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — (N)Gastrointestinal disorders * Colitis ulcerative * WORSENING OF ULCERATIVE COLITIS
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Group (N=16) | Low Dose Group (N=17) | Placebo (N=18)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 5 (5) | 3 (3) — Colitis ulcerative
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) — Abdominal pain
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) — Nausea
Dyspesia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) — Dyspesia
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) — vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-03-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT02493712/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT02493712/SAP_001.pdf